CLINICAL TRIAL: NCT00214357
Title: The Effects of Mindfulness Training on School Staff Emotions, Attention, and Stress
Brief Title: The Effects of Mindfulness Training on School Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2004-1277
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-11

CONDITIONS: Teachers
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction

SUMMARY:
The primary research objective is to investigate psychological, behavioral, and physiological changes in school staff as a result of undergoing meditation and stress reduction training. Specifically, we hypothesize that school staff undergoing meditation and stress reduction training will show decreased emotional distress on self-report measures, increased sustained attention on a behavioral task, and decreased stress levels as indexed by salivary cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Staff from Madison, WI area elementary school

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Self-report; behavioral task; diurnal cortisol

SECONDARY OUTCOMES:
Self-report measures

CONTACTS AND LOCATIONS:
Overall Officials: Donal G MacCoon, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States